CLINICAL TRIAL: NCT05973344
Title: Understanding and Anticipating Therapeutic and ADverse Responses in Anti-cancer Immune Checkpoint Inhibition Towards a Better Therapeutic Management of Patients
Acronym: TADIG-P
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0189 (TADIG-P); 2022-A02237-36 (Other: ANSM)
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the value of blood biomarkers for the purpose of predicting irAE development in cancer patients treated with immune checkpoint inihibitors (ICI) alone or in combination with other treatments (chemotherapy, radiotherapy and targeted therapy).

Data and blood samples will be collected from participants at different time points as part of routine follow-up visits. Data and blood samples will be analysed. Analysis will include the characterization of immune cells by mass and flow cytometry.

DETAILED DESCRIPTION:
Advances in treating patients with immunotherapy have dramatically changed cancer morbidity and mortality. Immune checkpoint inhibitors (ICI), alone or combined with other treatments, are currently used both as standard of care or in experimental settings for various cancers. ICI treatment induces objective clinical responses in 20-40% of patients (varies by tumor type); however, this leaves a majority of patients that do not respond to ICI therapy. ICI drugs purposely release immune regulatory controls and consequently increase immune activities; however, this release also provokes a significant risk of immunerelated adverse events (irAEs) such as dermatitis, hepatitis, thyroiditis and colitis, and less frequently but clinically important, hypophysitis, myocarditis and pneumonia. While the incidence of irAE is highly variable and influenced by many factors, Phase I and II trials reported rates from 10% to 80% for any grade irAE while an irAE of grade 3 or higher was observed in 2.5% to 18% of subjects. Recently, Jing et al. demonstrated that 20% of patients receiving anti-PD-1/PD-L1 had at least one irAE by integrating real-world pharmacovigilance of 26 tumor types for a total of 18,706 patients. Presently, the specific immune mechanism(s) driving irAE are unknown and biomarkers that predict their onset, particularly high-grade irAE, are urgently needed. For this reason, we hypothesize that an in-depth characterization and comparisons of the cell subpopulations composing and interacting within the primary cancer lesions, the peripheral blood, and in the organs in which irAE arise could help to better understand but also predict the clinical therapeutic response or/and irAE in patients with advanced cancers treated with ICI.

The research is a non-interventional monocentric prospective study of humans for the development of biological and medical knowledge, in which the procedures are performed and the products used in the usual manner, without additional or unusual diagnostic, treatment or monitoring procedures. The study includes patients monitored for their cancer at CHU of Brest and treated using Immune Checkpoint Inhibitors. Data and peripheral blood (47mL) will be collected at different time points as part of routine follow-up visits for analysis. Analysis will include the characterization of immune cells by mass and flow cytometry.

ELIGIBILITY:
* Age ≥ 18 years old
* ECOG performance status ≤ 1
* Must have histologically or cytologically confirmed tumour, eligible for treatment with ICI as standard-of-care alone or in combination with another ICI, ICI with chemotherapy, ICI with radiotherapy, or ICI with targeted therapy with no restrictions on number of prior systemic therapies
* Adequate bone marrow function as defined below

  * Absolute neutrophil count ≥ 1500/µL or 1.5x109/L
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 100000/µL or 100x109/L
* Adequate liver function as defined below

  * Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome < 3xUNL is allowed
  * AST (SGOT)/ALT (SGPT) ≤ 3.0 x ULN
  * Alkaline phosphatase ≤ 3.3 x ULN
* Adequate renal function as defined below

  _- Creatinine ≤ 1.5 x UNL or creatinine clearance > 60 mL/min
* Patient monitored for their cancer at CHU of Brest
* Did not oppose for their samples and clinical data to be used for translational research
* Non-opposition form obtained prior to any study related procedure

Exclusion Criteria:

* Patient with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study
* Patient already receiving ICI
* Primary immunodeficiency and/or history of allogenic transplantation
* Current active infection
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection)
* Subject of guardianship (tutorship, curatorship)
* Active pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with tumors treated with ICI (anti-CTLA-4, anti-PD-1/PD-L1, LAG3, etc.) as standard-of-care, alone or in combination with other treatments (chemotherapy, radiotherapy and targeted therapy)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2030-02-09 (Estimated); Study Completion 2030-02-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of irAE over the duration of the patient's follow-up | 36 months
  Apparition of irAE is appreciated according the physician definition. The description and grading scales of irAE found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.

SECONDARY OUTCOMES:
Survival (PFS). | 36 months
  PFS is defined as the time from random assignment in the clinical trial to disease progression or death from any cause.
Survival (OS). | 36 months
  OS is defined as the time from random assignment in the clinical trial to death.
Tumor response according to the iRECIST criteria | 36 months
  A copy of the iRECIST can be downloaded from the Lancet Oncology web site: https://www.thelancet.com/journals/lanonc/article/PIIS1470-2045(17)30074-8/fulltext

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Auberger, Principal Investigator — CHU Brest
Locations (1):
- Brest University Hospital, Brest, France